CLINICAL TRIAL: NCT01808768
Title: To Assess the Impact of Ocular Allergy Treatment on Patients Using an Opthalmic Agent (or no Treatment) Versus Alcaftadine(Lastacaft™)
Brief Title: Ocular Allergy Treatment Practical Impact Trial
Acronym: (OAT-PIT)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Starx Research Center, LLC (Industry)
Responsible Party: Principal Investigator, Jayesh G. Kanuga, M.D., Medical Doctor, Starx Research Center, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID IIT- 000373
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-03

CONDITIONS: Allergic Conjunctivitis; Rhinoconjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — alcaftadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alcaftadine (Experimental): subject on any ocular allergy ophthalmic treatment or no treatment will be started on Alcaftadine 0.25%(study drug)- 1 drop each eye daily for 1-2 weeks
  Interventions: Drug: Alcaftadine

INTERVENTIONS:
Drug: Alcaftadine — Alcaftadine 0.25% one dorp each eye daily for 1-2 weeks.
  Other Names: Lastacaft

SUMMARY:
To study the impact of alcaftadine in patients treated with other opthalmic ocular agents (or specific topical opthalmic treatment) in an allergy subspecialist outpatient setting.

DETAILED DESCRIPTION:
To assess the impact of ocular allergy treatment on patients using an ophthalmic agent (or no treatment) versus alcaftadine(Lastacaft™)

ELIGIBILITY:
Inclusion Criteria:

1. patients age 18 and older with a history of seasonal or perennial forms of allergic conjunctivitis and skin test positive reactivity to seasonal aeroallergens
2. Total Ocular Symptom Score (TOSS) on the day of enrollment of 4 or more.
3. have allergic ocular symptoms for the past week for which they are either treating with ophthalmic agents or have had no treatment.
4. Are willing/able to follow instructions from the study investigator and his/her study staff.
5. Have signed infromed consent approved by Institutional Review Board or Independent Ethics Committee.

   -

Exclusion Criteria:

1. Active ocular infection;
2. History of retinal detachment, diabetic neuropathy, or any progressive retinal disease;
3. Ocular surgical intervention within three (3) months prior to visit 1 or scheduled during the study.
4. History of unstable, or uncontrolled disease of any nature.
5. Pregnancy or lactation;
6. Have a known hypersensitivity tp LASTACAFT™ (alcaftadine) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Quality of Life- Eye Allergy Patient Impact Questionnaire | 4 months

SECONDARY OUTCOMES:
Ocular Surface Disease Index Pollen Count correlation of symptoms | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jayesh Kanuga, MD, Principal Investigator — Starx Research Center, LLC
Locations (2):
- United States (2):
  - STARx Research Center, Edison, New Jersey
  - STARx, Springfield, New Jersey